CLINICAL TRIAL: NCT06504355
Title: Enhancing Functional Fitness of Disabled Workers in Sheltered Workshops Through a Training Program Incorporating Resistive Action Video Games
Brief Title: Resistive Action Video Games Enhance Functional Fitness of Disabled Workers in Sheltered Workshops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Jen-Suh Chern, Associate Professor, National Taiwan Normal University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NSTC 110-2410-H-003 -109 -MY2
Record Dates: First submitted 2024-06-27; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Mental Disorder
Keywords: Disabled workers; Sheltered workshops; Functional fitness; Physical activities; Resistive video games; Action video games
MeSH Terms: conditions — Mental Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group participated in three 60-minute training sessions each week for 12 weeks. One of the session was group training. The other two session were individual training. In the group training session, the participants participate in the video aerobic exercise; in the individual sessions, the participants play action and resistive action video games: Fitness Boxing 2 and Adventure Ring-Fit. All participants in the experimental group wore a hear rate monitoring watch so that the researchers make sure that medium level of physical activities was achieved in each session. The participants underwent pre-, mid- and post-training measures of the outcome parameters which includes body weight, body mass index, basal metabolic rate, skeletal muscle rate, body fat percentage, flexibility, balance and agility.
  Interventions: Behavioral: Training program incorporating video aerobic exercise, action video game and resistive action video game
- Control group (No Intervention): The participants in the control group underwent no any special training but maintain daily work and leisure routines. They underwent pre-, mid- and post-experimental measures of the outcome parameters which was the same as those measured in the experimental group.

INTERVENTIONS:
Behavioral: Training program incorporating video aerobic exercise, action video game and resistive action video game — Participants in the experimental group participated in three 60-minute training sessions each week for 12 weeks. One of the session was group training. The other two session were individual training. In the group training session, the participants participate in the video aerobic exercise; in the individual sessions, the participants play action and resistive action video games: Fitness Boxing 2 and Adventure Ring-Fit. All participants in the experimental group wore a hear rate monitoring watch so that the researchers make sure that medium level of physical activities was achieved in each session.
  Arms: Experimental group

SUMMARY:
Aims: Investigating the efficacy of resistive action video games on functional fitness (FF) of disabled workers in sheltered workshops (DWSWs).

Methods: Thirty-two DWSWs participated in this study and were allocated as either experimental group (EG) or control group (CG). DWSWs in EG underwent three 60-minute sessions each week for 12 weeks; those in CG maintained daily routine. The outcomes included all components FF and were measures at pre-, mid- and post-training.

DETAILED DESCRIPTION:
Purpose: To investigate the efficacy of a training program including resistive action video games on functional fitness (FF) of disabled workers in sheltered workshops (DWSWs).

Material and methods: Thirty-two DWSWs participated in this study and were allocated as either experimental group (EG) or control group (CG). DWSWs in EG underwent three 60-minute training sessions each week for 12 weeks. One of the session is group training and two of the sessions are individual session. In group session, the participants do aerobic exercise following a video which was launch by the health management ministry of city government. In the individual session, the participants play play two video games alternatively. The video games used are Fitness Boxing 2 and Adventure Ring-Fit. In addition to the training program, the participants in the EG maintain work and leisure routine in addition to the added training. The participants in the CG maintained daily work and leisure routine.The outcome measures included body mass index, body weight, body fat percentage, skeletal muscle rate, muscle strength, cardiopulmonary endurance, flexibility, balance and agility. All participants must be evaluated of the outcome measures at pre-, mid- and post-training time point.

ELIGIBILITY:
Inclusion Criteria:

* (1) aged more than 20 years; (2) diagnosis of an intellectual disability, autism, or a psychiatric disorder; (3) employed for at least 6 hours per day and five days a week in the sheltered workshop; (4) capable of following verbal instructions to enable outcome measurement and of participating in the training program; and (5) voluntary agreement to participate and signed the informed consent form

Exclusion Criteria:

* (1) advisement against performing moderate- to high-intensity physical activities by a physician and (2) physical limitations preventing independent walking or standing without an assistive device.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Body weight | One week before training, 6 weeks of training, 12 weeks of training.
  On the counter Omron four-point bluetooth transmission weight and body fat meter HBF 702T was used
Body mass index | One week before training, 6 weeks of training, 12 weeks of training.
  On the counter Omron four-point bluetooth transmission weight and body fat meter HBF 702T was used
Body fat percentage | One week before training, 6 weeks of training, 12 weeks of training.
  On the counter Omron four-point bluetooth transmission weight and body fat meter HBF 702T was used
Skeletal muscle rate | One week before training, 6 weeks of training, 12 weeks of training.
  On the counter Omron four-point bluetooth transmission weight and body fat meter HBF 702T was used
Muscle strength | One week before training, after 6 weeks of training, after 12 weeks of training.
  Bicep arm curl test
Muscle strength | One week before training, after 6 weeks of training, after 12 weeks of training.
  Counts of strand-up in the 30-second chair stand test.
Cardiopulmonary endurance | One week before training, 6 weeks of training, 12 weeks of training.
  Counts of steps in the 2-minute step test
Flexibility | One week before training, 6 weeks of training, 12 weeks of training.
  The distance in centimeters between two middle fingers in the Back scratch test.
Flexibility | One week before training, 6 weeks of training, 12 weeks of training.
  The distance in centimeters between the middle fingers and the big toe in sit and reach test.
Balance | One week before training, 6 weeks of training, 12 weeks of training.
  Seconds to maintain one-leg stance stability
Agility | One week before training, 6 weeks of training, 12 weeks of training.
  Timed-Up-and-Go test

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Suh Chern, PhD, Principal Investigator — National Taiwan Normal University
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the individual participant data with other researchers.